CLINICAL TRIAL: NCT06939062
Title: Efficacy and Safety of Bipolar Resection Versus Enucleation of the Prostate in Management of Benign Prostatic Hyperplasia Patients With Medium-sized Prostates: A Prospective Randomized Controlled Clinical Trial
Brief Title: B-TURP vs BipolEP in Management of BPH Patients With Medium-sized Prostates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Atef Abdelaziz Mostafa, Lecturer of Urology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-TURP vs BipolEP
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia (BPH); Bipolar enucleation of the prostate (BipolEP); Bipolar Transurethral reaction of the prostate (B-TURP)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar enucleation of the prostate (BipolEP) patients (Active Comparator): Benign prostatic hyperplasia patients with medium -sized prostates who will undergo Bipolar enucleation of the prostate (BipolEP)
  Interventions: Procedure: Bipolar enucleation of the prostate (BipolEP)
- Bipolar transurethral resection of the prostate (B-TURP) patients (Active Comparator): Benign prostatic hyperplasia patients with medium -sized prostates who will undergo Bipolar transurethral resection of the prostate (B-TURP)
  Interventions: Procedure: Bipolar transurethral resection of the prostate (B-TURP)

INTERVENTIONS:
Procedure: Bipolar enucleation of the prostate (BipolEP) — Endoscopic transurethral enucleation of the prostate using bipolar energy
  Arms: Bipolar enucleation of the prostate (BipolEP) patients
Procedure: Bipolar transurethral resection of the prostate (B-TURP) — Endoscopic transurethral resection of the prostate using bipolar energy
  Arms: Bipolar transurethral resection of the prostate (B-TURP) patients

SUMMARY:
This is a comparative study of the efficacy and safety of endoscopic bipolar transurethral resection and enucleation of the prostate in management of benign prostatic hyperplasia patients with medium-sized prostates

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a highly prevalent condition among aging males, with incidence rates escalating progressively with age. Epidemiological data indicate that approximately 8% of men in their fourth decade are affected, a proportion that rises to 50% by the sixth decade and exceeds 80% in individuals reaching their ninth decade. BPH may induce bladder outlet obstruction (BOO), leading to lower urinary tract symptoms (LUTS). LUTS are one of the most frequent urological complaints in aging males. LUTS are typically categorized into obstructive and storage subtypes, with clinical BPH representing the predominant underlying etiology.

Approximately 20% of men with BPH will eventually require surgical intervention. Transurethral resection of the prostate (TURP) remains the gold-standard surgical treatment, offering both immediate relief of intravesical obstruction and durable improvement in voiding parameters and symptoms. However, the procedure carries significant risks, including perioperative bleeding and transurethral resection syndrome (TUR syndrome), with complication rates increasing proportionally to prostate size.

The recent technological advancements in urological equipment have led to increased adoption of bipolar transurethral resection of the prostate (B-TURP) for BPH management. This technique employs a plasma kinetic system that provides superior coagulation capabilities. A significant advantage of B-TURP is its use of normal saline irrigation, which substantially reduces the risk of TUR syndrome compared to conventional methods. Clinical studies have demonstrated B-TURP's efficacy in relieving bladder outlet obstruction secondary to BPH, with outcomes comparable to traditional approaches.

Despite advancements in TURP technology, incidence of complications such as postoperative recurrence remained unchanged, necessitating surgical innovation. In this context, bipolar enucleation of the prostate (BipoLEP) has emerged as an alternative technique designed to address these challenges. Our study was designed to conduct a comparative analysis of BipoLEP versus bipolar B-TURP in the treatment of medium-sized BPH patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 45-80 years with symptomatic BPH (IPSS ≥8).
* Prostate volume between 40-80 cc as determined by transrectal ultrasound (TRUS).
* Failure of medical management.
* Written informed consent.

Exclusion Criteria:

* Prostate cancer (suspected on PSA/DRE or confirmed by biopsy).
* Previous prostate/urethral surgery.
* Neurogenic bladder or urethral strictures.
* Significant coagulopathy.
* Uncontrolled urinary tract infection.
* Patient on anticoagulant medication.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in international prostate symptom score (IPSS) | At 6 months after the procedure (BipolEP or B-TURP)
  Treatment efficacy will be evaluated by comparing the change in international prostate symptom score (IPSS) between the two groups

SECONDARY OUTCOMES:
Complications | At 6 months after the procedure (BipolEP or B-TURP)
  Treatment safety will be evaluated by collecting and analyzing any reported complication within the first 6 postoperative months. Complications will be reported using the modified Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Urology Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to protect privacy of patients

REFERENCES:
- [Background] Chen S, Zhu L, Cai J, Zheng Z, Ge R, Wu M, Deng Z, Zhou H, Yang S, Wu W, Liao L, Tan J. Plasmakinetic enucleation of the prostate compared with open prostatectomy for prostates larger than 100 grams: a randomized noninferiority controlled trial with long-term results at 6 years. Eur Urol. 2014 Aug;66(2):284-91. doi: 10.1016/j.eururo.2014.01.010. Epub 2014 Jan 24. PMID 24502959
- [Background] Bhansali M, Patankar S, Dobhada S, Khaladkar S. Management of large (>60 g) prostate gland: PlasmaKinetic Superpulse (bipolar) versus conventional (monopolar) transurethral resection of the prostate. J Endourol. 2009 Jan;23(1):141-5. doi: 10.1089/end.2007.0005. PMID 19178175
- [Background] Ho HS, Yip SK, Lim KB, Fook S, Foo KT, Cheng CW. A prospective randomized study comparing monopolar and bipolar transurethral resection of prostate using transurethral resection in saline (TURIS) system. Eur Urol. 2007 Aug;52(2):517-22. doi: 10.1016/j.eururo.2007.03.038. Epub 2007 Mar 28. PMID 17416453
- [Background] Singh H, Desai MR, Shrivastav P, Vani K. Bipolar versus monopolar transurethral resection of prostate: randomized controlled study. J Endourol. 2005 Apr;19(3):333-8. doi: 10.1089/end.2005.19.333. PMID 15865523
- [Background] Ahyai SA, Gilling P, Kaplan SA, Kuntz RM, Madersbacher S, Montorsi F, Speakman MJ, Stief CG. Meta-analysis of functional outcomes and complications following transurethral procedures for lower urinary tract symptoms resulting from benign prostatic enlargement. Eur Urol. 2010 Sep;58(3):384-97. doi: 10.1016/j.eururo.2010.06.005. Epub 2010 Jun 11. PMID 20825758
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Kok ET, Schouten BW, Bohnen AM, Groeneveld FP, Thomas S, Bosch JL. Risk factors for lower urinary tract symptoms suggestive of benign prostatic hyperplasia in a community based population of healthy aging men: the Krimpen Study. J Urol. 2009 Feb;181(2):710-6. doi: 10.1016/j.juro.2008.10.025. Epub 2008 Dec 16. PMID 19091352
- [Background] GBD 2019 Benign Prostatic Hyperplasia Collaborators. The global, regional, and national burden of benign prostatic hyperplasia in 204 countries and territories from 2000 to 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Healthy Longev. 2022 Nov;3(11):e754-e776. doi: 10.1016/S2666-7568(22)00213-6. Epub 2022 Oct 20. PMID 36273485